CLINICAL TRIAL: NCT03655327
Title: Assessment of Upper Limb Joints Position During Reach and Grasp Functions in Different Heights and Weights in Sub-acute Stroke Patients
Brief Title: Reach to Grasp Movement of Stroke Patients: Different Heights and Weights
Status: Completed | Type: Observational
Sponsor: Ben-Gurion University of the Negev (Other)
Collaborators: Barzilai Medical Center (Other); Bet Hadar (Unknown)
Responsible Party: Principal Investigator, Shelly Levy-Tzedek, Assistant Professor, Ben-Gurion University of the Negev
Other Study IDs: 0014-17-BRZ
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Upper Extremity Paresis; Motor Control
Keywords: stroke rehabilitation
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stroke patients: stroke patients with upper limb paresis
  Interventions: Other: reach to grasp a cup
- healthy control group: healthy participants with no motor disability of the upper limb
  Interventions: Other: reach to grasp a cup

INTERVENTIONS:
Other: reach to grasp a cup — reach to grasp a cup of different weights located at different heights of table

SUMMARY:
A cross-sectional study of Reach-to-Grasp (RTG) movement of the upper limb of stroke patients vs. healthy controls. 30 stroke patients and 30 healthy controls will take place in a cross-sectional study. 3D kinematics and force regulation measures of RTG to a full and an empty cup at three different table heights will be measured. Motion analysis will include joint position and inter-limb coordination, velocity, and smoothness of movement. Data collected from the force sensor embaded in the cup will include peak force, time to peak force and variability in force production.

DETAILED DESCRIPTION:
Introduction Up to 75% of stroke survivors suffer persistent UL sensorimotor impairments, which considerably affect their ability to reach, pick up, and hold on to objects. Such deficits dramatically reduce the independence and, consequently, the quality of life, of post-stroke patients, and means for improving the effectiveness of post-stroke UL rehabilitation are much sought after. A prominent post-stoke UL impairment, which is strongly correlated with the level of the general post-stoke impairment and considerably affects daily activities and independence, is an impairment in reach-to-grasp (RTG) movements. Specifically, following stroke, movements become less smooth, less accurate, and less efficient than those of healthy individuals. As a result of such impairments, compensatory movements emerge, whereby the movement goal is achieved using an abnormal muscle activation pattern-e.g., excessive trunk displacement and a frontal hand orientation for grasping-which can lead to pain and fatigue. Retraining the coordination of RTG movements is, therefore, a major goal of post-stroke rehabilitation.

Despite extensive studies of post-stroke RTG movements, information is limited on how the height and weight of objects affect the ability of the impaired UL to reach and hold on to these objects - two crucial abilities for performing daily activities. Previous studies have shown that the height of the target object affects post-stroke RTG movements-namely, when post-stroke patients reach to higher targets, they recruit excessive compensatory muscles in the impaired UL, take longer to reach the target, demonstrate increased endpoint error, shoulder flexion, and abduction range of motion, and activate different muscle patterns to stabilize their trunks-highlighting the need to consider the height of target objects when formulating intervention programs to improve post-stroke RTG movements. However, most available studies of post-stroke UL RTG movements employed virtual tasks, which cannot accurately represent the physical world; It has been shown that, in both in stroke survivors and healthy individuals, an RTG task in a virtual 2D environment is slower, shorter, less straight, less accurate, and involves smaller ranges of shoulder and elbow joint excursions than an RTG task in a real, physical environment. These findings and others stress the importance of using real, daily objects of different heights to characterize and treat post-stroke UL RTG movement impairments. In addition, moving the arm while holding an object requires the individual to (unconsciously) increase the grip force to prevent the object from sliding, which may be impaired in post-stroke patients. However, clinical practitioners typically employ designated tools to measure grip forces after stroke-e.g., a dynamometer or a Pinch,-Grip,-Lift-and-Hold apparatus-rather than daily objects. The investigators are not familiar with studies that test lifting everyday objects of different weights following a stroke. Therefore, the first aim of the proposed study is to characterize the RTG movements and the grasp forces of post-stroke patients, as compared with those of healthy control individuals, attempting to reach, grasp, and lift real, functional, daily objects placed at different heights and of different weights.

Aim: to identify key differences between the RTG movements of post-stroke patients and healthy controls toward real objects of different weights and placed at different heights.

Comprehensively characterize the quality and efficacy of task-oriented RTG movements of sub-acute post-stroke patients and of healthy individuals to real, functional objects of different weights, placed at different heights (vertical distance from the participant), using a motion-capture system and a force sensor. Each participant repeats a RTG movement 18 times, 3 times each height and condition of cup (empty or full).

A total of 60 participants will take part in this study. Thirty hospitalized post-stroke patients will be recruited from the inpatient population of "Bet Hadar" geriatric rehabilitation center. In addition, thirty age-matched healthy control participans will be recruited from the community.

Procedure All participants will be examined individually by a single physical therapist (a master's student), in two 1-hour sessions. Evaluation of the control group will be performed in one session, lasting approximately 45 minutes. Stroke patients will be examined between one to two weeks before their discharge date from the rehabilitation center (average duration of rehabilitation in the hospital is two to three months). Stroke patients' measurement will be conducted in two separate days, in order to avoid fatigue, as it comprises both kinematic measurements and clinical mesurements.

The measurement session will be performed while the participants are in a sitting position, without back support, in front of a height-adjustable table. Participants will be instructed, once they hear a "beep" sound, to reach their hand at a self-selected speed, forward, toward a cup located on the table, lift it and place it on top of a five-centimeters-high block, positioned nearby. The participants will be instructed at the beginning of the session to avoid bending the trunk as much as possible during the reach movement, but no restraint of the trunk will be applied. The reach will be performed at three different heights: (a) low height- the height of the wrist when the hand is extended downwards, (b) medium height, ~75 cm from the floor, the height of a standard table and (c) high height- the height of the shoulder. The cup will be placed at an arm's distance, measured from the latral acromion to the radial styloid process, to avoid excessive trunk movement during the reach movement. This task was chosen as this is a functional everyday task.

In order to emphasize the everyday functionality of the task, in addition to the height variability, reach and grasp movements will be executed using a cup of two different weights: an empty cup and a cup full with water (250 ml). Participants will be informed whether the cup is full or empty. Lifting a cup primarily requires movement of the arm rather than the fingers. Hence, the role of the grasp is to stabilize the object and prevent undesirable movement. The reach will be executed by the affected arm of the post-stroke patients. Since the affected arm can be either their dominant or their non-dominant arm, the control group will be matched for dominance. That is, if half the patient group will reach with their non-dominant arm, then half of the control group will also be asked to reach with their non-dominant arm. Starting position for the low height will be with the arm held verticaly at the side of the body. Starting position for the medium and high heights will be with the arm placed on the ipsilateral thigh with palm facing down. Every reach combination of height and weight will be evaluated three times, according to the participant's ability. That is, while the maximal total number of reaching trials will be 18, some participants may not be able to complete all trials, due to arm weakness, fatigue, pain, etc. The order of the heights and weights will be set randomly using a computer program to prevent the influence of fatigue on one of the heights or weights.

Equipment Motion capture system: Position of the upper extremity joints during reach movements will be recorded by a motion capture system V120:Trio (OptiTrack, NaturalPoint, Inc., OR, USA) using eleven reflective markers placed on the participants' upper body. The V120:Trio tracking system is a portable multiple-camera, 6DoF optical object tracking technology. No calibration of the Trio system is required. Markers will be placed as follows: two markers will be placed vertically alligned on the sternum, to reflect the trunk motion, and one marker will be placed on each of the following anatomical landmarks: the lateral portion of the acromion-reflect the scapular motion, the proximal humerus, the lateral epicondyle of the elbow, the middle forearm, radial and ulnar styloid processes, the dorsal side of the palm at the axis along the middle part of the third metacarpal bone - to reflect the wrist motion, the index finger and the thumb. Additional two stationary vertical markers will be placed on the wall as reference points, and three additional markers will be placed on the cup and defined by the system as a rigid body. Data sampling speed of the Trio system is 120 Hz.

Force Sensor: Grip forces will be measured with a 3D force sensor (Nano25-E Transducer, ATI Industrial Automation, INC) embedded in the custom-built 3d-printed cup (see figure 3 in Appendix 1). The data sample speed of the force sensor is 100 Hz. Calibration of the sensor force is needed prior to every measurement trial (each reach movement). The data collected from the force sensor is the summed grip force applied on the cup.

ELIGIBILITY:
Inclusion Criteria:

1. First unilateral (ischemic or hemorrhagic) stroke with diagnosis confirmed by imaging from hospital discharge records.
2. Age 30-85 years.
3. Mini-Mental State Examination score ≥ 24/30.
4. Fugl-Meyer Upper Extremity score 16-66.
5. Pain level ≤ 4 on a 10-point Visual Analogue Scale.
6. Upper limb muscle tone assessed by Modified Ashworth Scale ≤ 2
7. Brunnstrom stages of motor recovery ≥ 3/7
8. Ability to sit independently without external support.

Exclusion Criteria:

1. Additional neurological problems (such us Parkinson's disease, unilateral neglect, pusher syndrome and apraxia).
2. Musculoskeletal, vision or sensory deficits affecting upper limb movements.
3. Aphasia affecting understanding of simple instructions.

   -

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: group 1: stroke patients with upper limb paresis group 2: healthy controls
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Index of curvature | 30 minutes
  the ratio between a straight line and the path of the movement the participant did

CONTACTS AND LOCATIONS:
Overall Officials: Ron Milo, MD, Principal Investigator — Barzilai Medical Center
Locations (1):
- Beit Hadar Geriatric center, Ashdod, South, Israel

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided. will be decided after data analysis